CLINICAL TRIAL: NCT03470727
Title: The Effect of Citrate Dialysate on Clot Formation and Anemia in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangkok Metropolitan Administration Medical College and Vajira Hospital (Other Government)
Responsible Party: Principal Investigator, Thananda Trakarnvanich, Associate Professor, Bangkok Metropolitan Administration Medical College and Vajira Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 71/2560
Record Dates: First submitted 2018-03-07; First posted 2018-03-20 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Hemodialysis; Citrate; Heparin

STUDY DESIGN:
Intervention Model Description: prospective comparison study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Citrate arm (Experimental): Citrate dialysate Phase 1 : Reduce heparin to 50% Phase 2: Reduce heparin to 25% Phase 3: Heparin free
  Interventions: Device: Citrate dialysate

INTERVENTIONS:
Device: Citrate dialysate — Change form acetate to citrate dialysate

SUMMARY:
Acetate-free citrate containing dialysate is expected to be clinically effective in maintaining hemodynamic stability during hemodialysis (HD). It has been demonstrated that citrate dialysate help produce a local anticoagulant effect by chelating ionized calcium. Moreover, citrate can improve phosphate and beta2 macroglobulin and better control of arterial hypertension and hemoglobinemia. We therefore would like to study the effect of citrate dialysate on clot formation and anemia while reducing heparin in chronic hemodialysis patients.

DETAILED DESCRIPTION:
This is the prospective comparison study. This study enrolled chronic hemodialysis patients age more than 18 who undergo hemodialysis 3 times per week for at least 3 months. All the patients should have serum ferritin 200-1000 ng/L and TSAT of 15-50%. The investigators exclude patients with age more than 70 years, comorbidities influencing citrate metabolism (hepatic failure,liver transplantation,cancer with bone metastasis), patients using heparin free protocol, hyperkalemia worsened by hypocalcemia, contraindication to heparin, treatment with cinacalcet or oral anticoagulant, patients using central venous catheter with blood flow less than 300 ml/min, and patients using low molecular weight heparin.

The study will be conducted in three phases over a period of 4 months. After run-in period for 2 weeks using acetate dialysate, the heparin dose will be titrated to lowest effective dose. During the first phase, citrate was replaced for acetate and heparin will be reduced to 50%. The second and third phase will be performed by reducing heparin doses to 25 % and heparin free consecutively. Each phase lasts for 4 weeks. Washout period for 2 weeks will be alternated after each phase.

Data collection: The investigators measure blood chemistries such as CBC, BUN creatinine electrolytes calcium phosphorus and KT/V at the beginning and at the end of each session. Ionized calcium will be monitored pre and post dialysis in each session. In addition, the investigators record clot score and erythropoietin dosage in each session and each phase.

ELIGIBILITY:
Inclusion Criteria:

* This study enrolled chronic hemodialysis patients age more than 18 who undergo hemodialysis 3 times per week for at least 3 months.
* Serum ferritin 200-1000 ng/L and TSAT of 15-50%.

Exclusion Criteria:

* age more than 70 years,
* comorbidities influencing citrate metabolism (hepatic failure,liver transplantation,cancer with bone metastasis),
* patients using heparin free protocol,hyperkalemia worsened by hypocalcemia
* contraindication to heparin,
* treatment with cinacalcet, or oral anticoagulant
* patients using central venous catheter with blood flow less than 300 ml/min
* patients using low molecular weight heparin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Effect of citrate dialysate to anemia | 3 months
  Hemoglobin in gram per dL

SECONDARY OUTCOMES:
Effect of citrate dialysate to dialyzer clotting | 3 months
  clot score.The clot score ranges from 1-4.Score 1 means no residual blood or less than 10 % in the fibers Score 2 means residual blood in < 10-25% of the fiber score 3 means residual blood in 25-50 % of the fiber Score 4 means more than 50 % of the fiber Score3
effect of citrate dialysate to electrolyte changes | 3 months
  electrolyte in mmoll/L(Sodium,Potassium,Chloride and bicarbonate)
effect of citrate dialysate to dialysis adequacy | 3 months
  Kt/V

CONTACTS AND LOCATIONS:
Overall Officials: Thananda Trakarnvanich, MD, Principal Investigator — Faculty of Medicine,Vajira Hospital,Navamindradhiraj University
Locations (1):
- Faculty of Medicine ,Vajira hospital,Navamindradhiraj University, Bangkok, Thailand